CLINICAL TRIAL: NCT02464033
Title: Open Label Trial to Evaluate the Tolerability of a Combination Therapy Consisting of GAD-alum (Diamyd®), Etanercept and Vitamin D in Children and Adolescents Newly Diagnosed With Type 1 Diabetes
Brief Title: EDCR Study - Etanercept Diamyd Combination Regimen -Open Trial to Evaluate Safety in Children With Type 1 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnny Ludvigsson (Other Government)
Collaborators: Swedish Child Diabetes Foundation (Other); Ostergotland County Council, Sweden (Other); Diamyd Medical AB (Industry)
Responsible Party: Sponsor-Investigator, Johnny Ludvigsson, MD, PhD, Professor, Linkoeping University
Organization: Linkoeping University (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EDCR IIa
Record Dates: First submitted 2015-05-19; First posted 2015-06-08 (Estimated); Results first posted 2019-09-25 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diamyd; Diabetes; Juvenile Diabetes; Diabetes Type 1; Type 1 Diabetes; Autoimmune Diabetes; Insulin Dependent Diabetes; Type 1 Diabetes MellitusType 1 Diabetes Mellitus; rhGAD65; GAD65; GAD-Alum; Diabetes Mellitus; Diabetes mellitus Type 1; Glucose Metabolism Disorders; Metabolic Diseases; Vitamin D; Etanercept
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Glucose Metabolism Disorders; Metabolic Diseases | interventions — Vitamin D; Cholecalciferol; Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): All patients will from Day 1 receive 2 000 IU vitamin D per os per day during 15 months, and from Days 1-90 receive etanercept (Enbrel) injected subcutaneously 0.8 mg/kg body weight (max 50 mg) once a week, and receive 2 subcutaneous injections of 20 μg Diamyd in a prime-and-boost regimen on Days 30 and 60.
  Interventions: Drug: GAD-Alum; Drug: Vitamin D; Drug: Etanercept

INTERVENTIONS:
Drug: GAD-Alum — Recombinant Human Glutamic Acid Decarboxylase (rhGAD65)
  Other Names: Diamyd
Drug: Vitamin D
  Other Names: Cholecalciferol
Drug: Etanercept

SUMMARY:
The objectives of this study is to:

* Evaluate the tolerability of a combination therapy with Diamyd, vitamin D and etanercept
* Evaluate how the above mentioned treatments influence the immune system and endogenous insulin secretion

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent given by patients and parent(s)/legal guardian(s)
2. Type 1 diabetes according to the ADA classification, diagnosed within the previous 100 days at the time of screening
3. Age 8.00 -17.99 years at time of screening
4. Fasting C-peptide at time of screening ≥0.12 nmol/L
5. Positive for GADA but < 50 000 Units
6. Menarchal females must agree to avoid pregnancy and have a negative urine pregnancy test
7. Immunity against Varicella, either through previous infection or vaccination
8. Patients must follow the Swedish vaccination programme
9. Patients of childbearing potential must agree to using adequate contraception, if sexually active, until 1 year after the last administration of GAD-alum and etanercept. Adequate contraception is as follows:

For females of childbearing potential:

1. oral (except low-dose gestagen (lynestrenol and norethisterone), injectable, or implanted hormonal contraceptives (females)
2. intrauterine device (females)
3. intrauterine system (for example, progestin-releasing coil) (females)
4. vasectomized male (with appropriate postvasectomy documentation of the absence of sperm in the ejaculate)

For males of childbearing potential:

a. Condom (male)

Exclusion Criteria:

1. Previous or current treatment with immunosuppressant therapy (although topical or inhaled steroids are accepted)
2. Continuous treatment with anti-inflammatory drug (sporadic treatment e.g. because of headache or in connection with fever a few days will be accepted)
3. Treatment with any oral or injected anti-diabetic medications (especially hypoglycemic agents) other than insulin
4. Treatment with Vitamin D, marketed or not, or unwilling to abstain from such medication during the trial
5. A history of hypercalcemia
6. A history of anaemia or significantly abnormal haematology results at screening
7. A history of epilepsy, head trauma or cerebro-vascular accident, or clinical features of continuous motor unit activity in proximal muscles
8. Clinically significant history of acute reaction to vaccines or other drugs in the past
9. Treatment with any vaccine within 4 months prior to planned first administration of GAD-Alum or planned treatment with vaccine up to 4 months after the last injection with GAD-Alum, including influenza vaccine
10. Participation in other clinical trials with a new chemical entity within the previous 3 months
11. Inability or unwillingness to comply with the provisions of this protocol
12. A history of alcohol or drug abuse
13. A significant illness other than diabetes within 2 weeks prior to first dosing
14. Known human immunodeficiency virus (HIV)
15. Prior or active viral hepatitis B or C infection
16. Females who are lactating or pregnant (for females who have started menstruating the possibility of pregnancy must be excluded by urine βHCG on-site within 24 hours prior to the GAD-Alum and etanercept administration, respectively)
17. Males or females not willing to use adequate contraception, if sexually active, until 1 year after the last GAD-Alum and etanercept administration, respectively
18. Presence of associated serious disease or condition, including active skin infections that preclude subcutaneous injection, which in the opinion of the investigator makes the patient non-eligible for the study.
19. Deemed by the investigator not being able to follow instructions and/or follow the study protocol
20. Active infection, including chronic and local infection or a history of previous tendency to serious infections, recent or ongoing uncontrolled bacterial, viral, fungal or other opportunistic infections, or known infection with active EBV or CMV
21. Hypersensitivity to the active substance in Enbrel (etanercept) or other ingredients in Enbrel
22. Active or inactive (latent) tuberculosis (TBC) at screening
23. History of malignancy or significant cardiovascular disease
24. Current or history of leukopenia, anemia and/or thrombocytopenia
25. Liver disease (clinical or hepatic enzymes >3 times the upper limit of normal (ULN))
26. Renal insufficiency (clinical or creatinine >3 times the upper limit of normal (ULN))
27. MS, undefined neurologic condition or known SLE, or anti-nuclear or known doublestranded DNA antibody positivity
28. Arrhythmia
29. Pancreatitis
30. Vitamin D serum levels >100 nmol/L at screening

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2015-05; Primary Completion 2019-02-25 (Actual); Study Completion 2019-02-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnny Ludvigsson, MD,PhD,Prof, Principal Investigator — Linkoeping University
Locations (8):
- Sweden (8):
  - Helsingborg Hospital, Helsingborg
  - Linköping University Hospital, Linköping
  - Lund University Hospital, Lund
  - Skåne University Hospital, UMAS, Malmo
  - Örebro University Hospital, Örebro
  - Sachsska, Södersjukhuset, Stockholm
  - Uddevalla Hospital, Uddevalla
  - Västerås Hospital, Västerås

RESULTS

PARTICIPANT FLOW:
Groups:
- GAD-Alum+Vitamin D+Etanercept: All patients will from Day 1 receive 2000 IU vitamin D per os per day during 15 months, and from Days 1-90 receive etanercept (Enbrel) injected subcutaneously 0.8 mg/kg body weight (max 50 mg) once a week, and receive 2 subcutaneous injections of 20 μg Diamyd in a prime-and-boost regimen on Days 30 and 60.
  GAD-Alum
  Vitamin D
  Etanercept
Period: Overall Study
Arm/Group | GAD-Alum+Vitamin D+Etanercept
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- GAD-Alum+Vitamin D+Etanercept: All patients will from Day 1 receive 2 000 IU vitamin D per os per day during 15 months, and from Days 1-90 receive etanercept (Enbrel) injected subcutaneously 0.8 mg/kg body weight (max 50 mg) once a week, and receive 2 subcutaneous injections of 20 μg Diamyd in a prime-and-boost regimen on Days 30 and 60.
  GAD-Alum
  Vitamin D
  Etanercept
Arm/Group | GAD-Alum+Vitamin D+Etanercept
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.36 (2.321)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Sweden | 20
Type 1 Diabetes duration [Mean (Standard Deviation); unit: days] | 81.35 (22.091)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 18.38 (2.141)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Reactions of the Injection Site as an Assessment of the Tolerability
Description: Number of patients with reactions of the injection site (Erythema, Oedema, Haematoma, Tenderness, Pain, Itching, Other). Inspection of injection site 60 minutes after GAD-Alum injection by investigator or nurse
Time Frame: 1 months
Population: Safety
Measure: Count of Participants; unit: Participants
Arm/Group | GAD-Alum+Vitamin D+Etanercept
Number analyzed (Participants) | 20
Participants | 3

2. Primary Outcome: Number of Patients With Reactions of the Injection Site as an Assessment of the Tolerability
Description: as for outcome 1
Time Frame: 2 months
Population: Safety
Measure: Count of Participants; unit: Participants
Arm/Group | GAD-Alum+Vitamin D+Etanercept
Number analyzed (Participants) | 20
Participants | 5

3. Primary Outcome: Number of Patients With Any Abnormal Findings From Physical Examinations After Baseline
Description: Number of patients with any abnormal findings from physical examinations after baseline, including neurological assessments as an assessment of tolerability.
Time Frame: Month 1, 2, 3, 6, 9, 15 and 30
Population: Safety
Measure: Count of Participants; unit: Participants
Arm/Group | GAD-Alum+Vitamin D+Etanercept
Number analyzed (Participants) | 20
Participants | 6

4. Primary Outcome: Number of Patients With Clinically Significant Laboratory Findings
Description: Number of patients with clinically significant laboratory findings, laboratory measurements as an assessment of the tolerability
Time Frame: Month 1, 2, 3, 6, 9, 15 and 30
Population: Safety
Measure: Count of Participants; unit: Participants
Arm/Group | GAD-Alum+Vitamin D+Etanercept
Number analyzed (Participants) | 20
Participants | 0

5. Primary Outcome: GAD65AB Titer Measured to Evaluate the Tolerability (Main Study Period)
Description: GAD65AB titer (GADA) change from baseline. GAD65AB = Antibodies to GAD with molecular mass 65000
Time Frame: 6 months
Population: Intention To Treat (ITT)
Measure: Mean (Standard Deviation); unit: U/mL
Arm/Group | GAD-Alum+Vitamin D+Etanercept
Number analyzed (Participants) | 20
U/mL | 2509.41 (4866.515)

6. Primary Outcome: GAD65AB Titer Measured to Evaluate the Tolerability (Main Study Period)
Description: GAD65AB titer (GADA) change from baseline. GAD65AB = Antibodies to GAD with molecular mass 65000
Time Frame: 15 months
Population: ITT
Measure: Mean (Standard Deviation); unit: U/mL
Arm/Group | GAD-Alum+Vitamin D+Etanercept
Number analyzed (Participants) | 20
U/mL | 1036.19 (2527.249)

7. Primary Outcome: GAD65AB Titer Measured to Evaluate the Tolerability (Main Study Period)
Description: GAD65AB titer (GADA) change from baseline. GAD65AB = Antibodies to GAD with molecular mass 65000
Time Frame: 30 months
Population: ITT
Measure: Mean (Standard Deviation); unit: U/mL
Arm/Group | GAD-Alum+Vitamin D+Etanercept
Number analyzed (Participants) | 20
U/mL | 347.01 (1564.466)

8. Primary Outcome: Number of Patients With an Infection Reported as Adverse Event Related to Study Treatment
Description: Number of patients with an infection reported as Adverse Event related to study treatment (GAD-Alum and/or Etanercept),as an assessment of the tolerability
Time Frame: Month 1, 2, 3, 6, 9, 15 and 30
Population: Safety
Measure: Count of Participants; unit: Participants
Arm/Group | GAD-Alum+Vitamin D+Etanercept
Number analyzed (Participants) | 20
Participants | 3

9. Secondary Outcome: C-peptide: Area Under the Curve (AUC 0-120 Min) During an MMTT, Change From Baseline
Description: Weighted mean C-peptide: (AUC mean 0-120 min) during an MMTT, change from baseline to 6 months. MMTT=Mixed Meal Tolerance Test
Time Frame: Baseline and 6 months at 0, 30, 60, 90 and 120 minutes post-dose
Population: ITT, MMTT not performed for 2 patients hence no data available for 2 out of the 20 patients
Measure: Mean (Standard Deviation); unit: nmol/L*min
Arm/Group | GAD-Alum+Vitamin D+Etanercept
Number analyzed (Participants) | 18
nmol/L*min | -0.09 (0.153)

10. Secondary Outcome: C-peptide: Area Under the Curve (AUC 0-120 Min) During an MMTT, Change From Baseline
Description: Weighted mean C-peptide: (AUC mean 0-120 min) during an MMTT, change from baseline to 15 months
Time Frame: Baseline and 15 months at 0, 30, 60, 90 and 120 minutes post-dose
Population: ITT
Measure: Mean (Standard Deviation); unit: nmol/L*min
Arm/Group | GAD-Alum+Vitamin D+Etanercept
Number analyzed (Participants) | 20
nmol/L*min | -0.30 (0.158)

11. Secondary Outcome: C-peptide: Area Under the Curve (AUC 0-120 Min) During an MMTT, Change From Baseline
Description: Weighted mean C-peptide: (AUC mean 0-120 min) during an MMTT, change from baseline to 30 months
Time Frame: Baseline and 30 months at 0, 30, 60, 90 and 120 minutes post-dose
Population: ITT, , MMTT not performed for 1 patient hence no data available for 1 out of the 20 patients
Measure: Mean (Standard Deviation); unit: nmol/L*min
Arm/Group | GAD-Alum+Vitamin D+Etanercept
Number analyzed (Participants) | 19
nmol/L*min | -0.40 (0.168)

12. Secondary Outcome: Number of Patients With a Stimulated Maximum C-peptide Level Above 0.2 Nmol/L
Description: Number of patients with a stimulated maximum C-peptide level above 0.2 nmol/L at 6 months
Time Frame: 6 months
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | GAD-Alum+Vitamin D+Etanercept
Number analyzed (Participants) | 20
Participants | 17

13. Secondary Outcome: Number of Patients With a Stimulated Maximum C-peptide Level Above 0.2 Nmol/L
Description: Number of patients with a stimulated maximum C-peptide level above 0.2 nmol/L at 15 months
Time Frame: 15 months
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | GAD-Alum+Vitamin D+Etanercept
Number analyzed (Participants) | 20
Participants | 14

14. Secondary Outcome: Number of Patients With a Stimulated Maximum C-peptide Level Above 0.2 Nmol/L
Description: Number of patients with a stimulated maximum C-peptide level above 0.2 nmol/L at 30 months
Time Frame: 30 months
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | GAD-Alum+Vitamin D+Etanercept
Number analyzed (Participants) | 20
Participants | 8

15. Secondary Outcome: Hemoglobin A1c (HbA1c), Change From Baseline
Description: Hemoglobin A1c (HbA1c), change from baseline to 6 months
Time Frame: Baseline and 6 months
Population: ITT
Measure: Mean (Standard Deviation); unit: mmol/mol
Arm/Group | GAD-Alum+Vitamin D+Etanercept
Number analyzed (Participants) | 20
mmol/mol | 0.80 (8.433)

16. Secondary Outcome: Hemoglobin A1c (HbA1c), Change From Baseline
Description: Hemoglobin A1c (HbA1c), change from baseline to 15 months
Time Frame: Baseline and 15 months
Population: ITT
Measure: Mean (Standard Deviation); unit: mmol/mol
Arm/Group | GAD-Alum+Vitamin D+Etanercept
Number analyzed (Participants) | 20
mmol/mol | 6.15 (12.495)

17. Secondary Outcome: Hemoglobin A1c (HbA1c), Change From Baseline
Description: Hemoglobin A1c (HbA1c), change from baseline to 30 months
Time Frame: Baseline and 30 months
Population: ITT
Measure: Mean (Standard Deviation); unit: mmol/mol
Arm/Group | GAD-Alum+Vitamin D+Etanercept
Number analyzed (Participants) | 20
mmol/mol | 7.55 (11.213)

18. Secondary Outcome: Exogenous Insulin Dose Per kg Body Weight and 24 Hours, Change From Baseline
Description: Exogenous 24-hour insulin dose per kg body weight and 24 hours average, change from baseline
Time Frame: Baseline and 6 months
Population: ITT
Measure: Mean (Standard Deviation); unit: IU
Arm/Group | GAD-Alum+Vitamin D+Etanercept
Number analyzed (Participants) | 20
IU | 0.01 (0.249)

19. Secondary Outcome: Exogenous Insulin Dose Per kg Body Weight and 24 Hours, Change From Baseline
Description: Exogenous 24-hour insulin dose per kg body weight and 24 hours average, change from baseline
Time Frame: Baseline and 15 months
Population: ITT
Measure: Mean (Standard Deviation); unit: IU
Arm/Group | GAD-Alum+Vitamin D+Etanercept
Number analyzed (Participants) | 20
IU | 0.25 (0.342)

20. Secondary Outcome: Exogenous Insulin Dose Per kg Body Weight and 24 Hours, Change From Baseline
Description: Exogenous 24-hour insulin dose per kg body weight and 24 hours average, change from baseline
Time Frame: Baseline and 30 months
Population: ITT
Measure: Mean (Standard Deviation); unit: IU
Arm/Group | GAD-Alum+Vitamin D+Etanercept
Number analyzed (Participants) | 20
IU | 0.42 (0.333)

21. Secondary Outcome: C-peptide: Stimulated, 90 Minute Value, Change From Baseline
Description: C-peptide: Stimulated, 90 minute value, change from baseline to 6 months
Time Frame: Baseline and 6 months
Population: ITT, not performed for 2 patients hence no data available for 2 out of the 20 patients
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | GAD-Alum+Vitamin D+Etanercept
Number analyzed (Participants) | 18
nmol/L | -0.09 (0.233)

22. Secondary Outcome: C-peptide: Stimulated, 90 Minute Value, Change From Baseline
Description: C-peptide: Stimulated, 90 minute value, change from baseline to 15 months
Time Frame: Baseline and 15 months
Population: ITT
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | GAD-Alum+Vitamin D+Etanercept
Number analyzed (Participants) | 20
nmol/L | -0.35 (0.231)

23. Secondary Outcome: C-peptide: Stimulated, 90 Minute Value, Change From Baseline
Description: C-peptide: Stimulated, 90 minute value, change from baseline to 30 months
Time Frame: Baseline and 30 months
Population: ITT, not performed for 1 patient hence no data available for 1 out of the 20 patients
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | GAD-Alum+Vitamin D+Etanercept
Number analyzed (Participants) | 19
nmol/L | -0.49 (0.221)

24. Secondary Outcome: C-peptide Fasting Concentration, Change From Baseline
Description: C-peptide: Fasting concentration, change from baseline to 6 months
Time Frame: Baseline and 6 months
Population: ITT
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | GAD-Alum+Vitamin D+Etanercept
Number analyzed (Participants) | 20
nmol/L | -0.02 (0.083)

25. Secondary Outcome: C-peptide Fasting Concentration, Change From Baseline
Description: C-peptide: Fasting, concentration, change from baseline to 15 months
Time Frame: Baseline and 15 months
Population: ITT
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | GAD-Alum+Vitamin D+Etanercept
Number analyzed (Participants) | 20
nmol/L | -0.10 (0.091)

26. Secondary Outcome: C-peptide Fasting Concentration, Change From Baseline
Description: C-peptide: Fasting, concentration, change from baseline to 30 months
Time Frame: Baseline and 30 months
Population: ITT
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | GAD-Alum+Vitamin D+Etanercept
Number analyzed (Participants) | 20
nmol/L | -0.15 (0.093)

27. Secondary Outcome: Spontaneous IL-17a Secretion
Description: Spontaneous IL-17a secretion at baseline, 6 months, 9 months, 15 months and 30 months
Time Frame: Baseline, 6 months, 9 months, 15 months and 30 months
Population: ITT
Measure: Median (Standard Deviation); unit: pg/ml
Arm/Group | GAD-Alum+Vitamin D+Etanercept
Number analyzed (Participants) | 20
pg/ml
  IL-17a, Baseline | 3.16 (8.36)
  IL-17a, 6 months: number analyzed (Participants) | 19
  IL-17a, 6 months | 6.07 (10.13)
  IL-17a, 9 months | 7.06 (11.35)
  IL-17a,15 months: number analyzed (Participants) | 18
  IL-17a,15 months | 6.54 (7.83)
  IL-17a, 30 months: number analyzed (Participants) | 18
  IL-17a, 30 months | 4.75 (10.64)

28. Secondary Outcome: GAD65-induced IL-4 Secretion
Description: GAD65-induced IL-4 secretion at baseline, 6 months, 9 months, 15 months, 30 months
Time Frame: Baseline, 6 months, 9 months, 15 months, 30 months
Population: ITT
Measure: Median (Standard Deviation); unit: pg/ml
Arm/Group | GAD-Alum+Vitamin D+Etanercept
Number analyzed (Participants) | 20
pg/ml
  IL-4, baseline | 0.01 (1.03)
  IL-4, 6 months | 0.01 (0.58)
  IL-4, 9 months: number analyzed (Participants) | 19
  IL-4, 9 months | 0.01 (1.21)
  IL-4, 15 months: number analyzed (Participants) | 18
  IL-4, 15 months | 0.01 (1.52)
  IL-4, 30 months: number analyzed (Participants) | 18
  IL-4, 30 months | 0.01 (0.63)

29. Secondary Outcome: GAD65-induced IL-13 Secretion
Description: GAD65-induced IL-13 secretion at baseline, 6 months, 9 months, 15 months, 30 months
Time Frame: Baseline, 6 months, 9 months, 15 months, 30 months
Population: ITT
Measure: Median (Standard Deviation); unit: pg/ml
Arm/Group | GAD-Alum+Vitamin D+Etanercept
Number analyzed (Participants) | 20
pg/ml
  IL-13, Baseline | 0.01 (56.88)
  IL-13, 6 months: number analyzed (Participants) | 19
  IL-13, 6 months | 1.67 (58.47)
  IL-13, 9 months | 5.12 (69.63)
  IL-13, 15 months: number analyzed (Participants) | 18
  IL-13, 15 months | 0.01 (99.00)
  IL-13, 30 months | 0.01 (49.95)

30. Secondary Outcome: GAD65-induced IFN-gamma Secretion
Description: GAD65-induced IFN-gamma secretion at baseline, 6 months, 9 months, 15 months, 30 months
Time Frame: Baseline, 6 months, 9 months, 15 months, 30 months
Population: ITT
Measure: Median (Standard Deviation); unit: pg/ml
Arm/Group | GAD-Alum+Vitamin D+Etanercept
Number analyzed (Participants) | 20
pg/ml
  IFN-gamma, baseline | 4.39 (210.52)
  IFN-gamma, 6 months: number analyzed (Participants) | 19
  IFN-gamma, 6 months | 11.44 (223.16)
  IFN-gamma, 9 months: number analyzed (Participants) | 19
  IFN-gamma, 9 months | 22.77 (679.35)
  IFN-gamma, 15 months: number analyzed (Participants) | 18
  IFN-gamma, 15 months | 0.01 (1679.59)
  IFN-gamma, 30 months: number analyzed (Participants) | 18
  IFN-gamma, 30 months | 0.01 (227.91)

31. Secondary Outcome: GAD65-induced TNF-alpha Secretion
Description: GAD65-induced TNF-alpha secretion at baseline, 6 months, 9 months, 15 months, 30 months
Time Frame: Baseline, 6 months, 9 months, 15 months, 30 months
Population: ITT
Measure: Median (Standard Deviation); unit: pg/ml
Arm/Group | GAD-Alum+Vitamin D+Etanercept
Number analyzed (Participants) | 20
pg/ml
  TNF-alpha, baseline | 0.01 (348.28)
  TNF-alpha, 6 months: number analyzed (Participants) | 19
  TNF-alpha, 6 months | 0.01 (89.19)
  TNF-alpha, 9 months: number analyzed (Participants) | 19
  TNF-alpha, 9 months | 0.01 (355.09)
  TNF-alpha, 15 months: number analyzed (Participants) | 18
  TNF-alpha, 15 months | 0.01 (362.35)
  TNF-alpha, 30 months: number analyzed (Participants) | 18
  TNF-alpha, 30 months | 0.01 (206.37)

32. Secondary Outcome: GAD65-induced GM-CSF Secretion
Description: GAD65-induced GM-CSF secretion baseline, 6 months, 9 months, 15 months, 30 months
Time Frame: Baseline, 6 months, 9 months, 15 months, 30 months
Population: ITT
Measure: Median (Standard Deviation); unit: pg/ml
Arm/Group | GAD-Alum+Vitamin D+Etanercept
Number analyzed (Participants) | 20
pg/ml
  GM-CSF, baseline | 0.01 (16.96)
  GM-CSF, 6 months: number analyzed (Participants) | 19
  GM-CSF, 6 months | 0.01 (18.00)
  GM-CSF, 9 months: number analyzed (Participants) | 19
  GM-CSF, 9 months | 1.52 (24.70)
  GM-CSF, 15 months: number analyzed (Participants) | 18
  GM-CSF, 15 months | 0.01 (36.95)
  GM-CSF, 30 months: number analyzed (Participants) | 18
  GM-CSF, 30 months | 0.01 (6.00)

33. Secondary Outcome: GAD65-induced MIP-1b Secretion
Description: GAD65-induced MIP-1b secretion at baseline, 6 months, 9 months, 15 months, 30 months
Time Frame: Baseline, 6 months, 9 months, 15 months, 30 months
Population: ITT
Measure: Median (Standard Deviation); unit: pg/ml
Arm/Group | GAD-Alum+Vitamin D+Etanercept
Number analyzed (Participants) | 20
pg/ml
  MIP-1b, baseline | 0.01 (85.46)
  MIP-1b, 6 months: number analyzed (Participants) | 19
  MIP-1b, 6 months | 0.01 (57.78)
  MIP-1b, 9 months: number analyzed (Participants) | 19
  MIP-1b, 9 months | 0.01 (134.30)
  MIP-1b, 15 months: number analyzed (Participants) | 18
  MIP-1b, 15 months | 30.64 (302.04)
  MIP-1b, 30 months: number analyzed (Participants) | 18
  MIP-1b, 30 months | 14.61 (72.54)

34. Secondary Outcome: GAD65-induced MCP-1 Secretion
Description: GAD65-induced MCP-1 secretion at baseline, 6 months, 9 months, 15 months, 30 months
Time Frame: Baseline, 6 months, 9 months, 15 months, 30 months
Population: ITT
Measure: Median (Standard Deviation); unit: pg/ml
Arm/Group | GAD-Alum+Vitamin D+Etanercept
Number analyzed (Participants) | 20
pg/ml
  MCP-1, baseline | 0.01 (106.61)
  MCP-1, 6 months: number analyzed (Participants) | 19
  MCP-1, 6 months | 38.54 (89.74)
  MCP-1, 9 months: number analyzed (Participants) | 19
  MCP-1, 9 months | 0.01 (144.03)
  MCP-1, 15 months: number analyzed (Participants) | 18
  MCP-1, 15 months | 24.42 (203.74)
  MCP-1, 30 months: number analyzed (Participants) | 18
  MCP-1, 30 months | 37.50 (220.66)

ADVERSE EVENTS:
Time Frame: 30 months
Description: Adverse Events were recorded in the Case Report Form at each clinic visit.
Arm/Group | GAD-Alum+Vitamin D+Etanercept
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 20/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GAD-Alum+Vitamin D+Etanercept (N=20)
Gastroenteritis (Infections and infestations) | 9 (11)
Influenza (Infections and infestations) | 2 (2)
Nasopharyngitis (Infections and infestations) | 13 (30)
Viral infection (Infections and infestations) | 8 (15)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2)
Depression (Psychiatric disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Injection site reaction (General disorders) | 13 (20)
Pyrexia (General disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-17): https://cdn.clinicaltrials.gov/large-docs/33/NCT02464033/Prot_SAP_000.pdf